CLINICAL TRIAL: NCT01805479
Title: Exercise Training in Depressed Traumatic Brain Injury Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants. Sponsor requested study closure.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PT107574; 7K23HD067553 (NIH)
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Traumatic Brain Injury
Keywords: exercise; depression; traumatic brain injury
MeSH Terms: conditions — Depression; Brain Injuries, Traumatic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stretching-flexibility (Placebo Comparator): This group will use a stretching and flexibility program designed to utilize minimal levels of aerobic capacity. It was chosen in place of a education-based control group due to the high level of personal interaction that is found in the active arm.
  Interventions: Other: stretching and flexibility program
- aerobic exercise group (Active Comparator): aerobic activity targeting 60% peak heart rate for 12 weeks is the active group.
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — the active arm will be asked to perform 60% of maximum heart rate
  Arms: aerobic exercise group
Other: stretching and flexibility program — stretching and flexibility program for the Placebo Comparator Arm
  Arms: stretching-flexibility

SUMMARY:
The purpose of this study is to determine the feasibility of successfully delivering moderate intensity aerobic exercise training to depressed traumatic brain injury subjects between one and three years after injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) alters the lives of many civilians and those involved in armed conflicts. Sequelae of TBI includes depression in up to 30% of cases. Appearance of depression after TBI impairs recovery and results in sub-optimal re-integration into society. Treatment of post TBI depression relies on oral medications, whose efficacy and side effect profile is sub-optimal. Exercise training is effective in spontaneous depression as a stand alone treatment and in conjunction with oral medications, and this may represent an alternative treatment option in the TBI population. Further, the pathophysiology of depression after TBI has yet to be examined with the full scientific rigor required. This project proposes to use exercise training of moderate intensity as a treatment for depression after TBI, while measuring biological markers as a way to investigate efficacy and provide insight into the pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* CT brain with subdural hematoma, subarachnoid hemorrhage, and/or cortical contusion
* Glasgow outcome scale extended of 4 to 8
* speaks English
* Beck Depression Inventory -II score between 14 and 28
* sedentary life style
* one to three years after traumatic brain injury

Exclusion Criteria:

* prior history of brain process (example, stroke, brain tumor)
* aphasia
* psychosis, mania, bipolar disorder, schizophrenia
* pregnancy
* inability to exercise via cycles or treadmill

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
completion of exercise protocol | 12 weeks
  The primary aim is to measure the rate of completion of the exercise protocol.

SECONDARY OUTCOMES:
neuropsychological testing | pre and post intervention, week zero and week 13
  cognitive testing battery will be performed to examine the impact of exercise on cognition in depressed traumatic brain injury subjects. Administered to both arms.
mood assessment | week 0, week 13, and weekly during 12 week intervention
  depression symptom inventories will be performed to examine the impact of exercise on cognition in depressed traumatic brain injury subjects. Administered to both arms.
Columbia-Suicide Severity Rating Scale | week 0, week 13, and weekly during 12 week intervention
  Columbia-Suicide Severity Rating Scale was developed to meet the need for tracking changes in a person's suicidal thinking and behavior over time, and to determine who is most at risk. Administered to both arms.
magnetic resonance imaging | week 0, week 13
  MRI will be done before and after exercise protocol on a subset of subjects. Selection of these subjects will be done by randomization, starting once the MRI is available for use. The purpose is to examine the brain for exercise influenced volumetric changes. Administered to a subset of both arms of the study.
biochemical assays | week 0, week 13
  brain-derived neurotrophic factor, vascular endothelial growth factor, insulin-like growth factor-1. The listed neurotrophic factors have been linked to depression and have been shown to be influenced by exercise. The impact of depression and exercise in the context of traumatic brain injury is unknown. Administered to both study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hudak, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. The DOSE study: a clinical trial to examine efficacy and dose response of exercise as treatment for depression. Control Clin Trials. 2002 Oct;23(5):584-603. doi: 10.1016/s0197-2456(02)00226-x. PMID 12392873
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. Exercise treatment for depression: efficacy and dose response. Am J Prev Med. 2005 Jan;28(1):1-8. doi: 10.1016/j.amepre.2004.09.003. PMID 15626549
- [Background] Hudak A, Warner M, Marquez de la Plata C, Moore C, Harper C, Diaz-Arrastia R. Brain morphometry changes and depressive symptoms after traumatic brain injury. Psychiatry Res. 2011 Mar 31;191(3):160-5. doi: 10.1016/j.pscychresns.2010.10.003. PMID 21310594
- [Background] Jorge RE, Robinson RG, Arndt SV, Starkstein SE, Forrester AW, Geisler F. Depression following traumatic brain injury: a 1 year longitudinal study. J Affect Disord. 1993 Apr;27(4):233-43. doi: 10.1016/0165-0327(93)90047-n. PMID 8509524
- [Background] Fann JR, Katon WJ, Uomoto JM, Esselman PC. Psychiatric disorders and functional disability in outpatients with traumatic brain injuries. Am J Psychiatry. 1995 Oct;152(10):1493-9. doi: 10.1176/ajp.152.10.1493. PMID 7573589
- [Background] van Reekum R, Bolago I, Finlayson MA, Garner S, Links PS. Psychiatric disorders after traumatic brain injury. Brain Inj. 1996 May;10(5):319-27. doi: 10.1080/026990596124340. PMID 8735663
- [Background] Gomez-Hernandez R, Max JE, Kosier T, Paradiso S, Robinson RG. Social impairment and depression after traumatic brain injury. Arch Phys Med Rehabil. 1997 Dec;78(12):1321-6. doi: 10.1016/s0003-9993(97)90304-x. PMID 9421985
- [Background] Rapoport MJ, Kiss A, Feinstein A. The impact of major depression on outcome following mild-to-moderate traumatic brain injury in older adults. J Affect Disord. 2006 Jun;92(2-3):273-6. doi: 10.1016/j.jad.2005.05.022. Epub 2006 Feb 28. PMID 16504305
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Silver JM, Kramer R, Greenwald S, Weissman M. The association between head injuries and psychiatric disorders: findings from the New Haven NIMH Epidemiologic Catchment Area Study. Brain Inj. 2001 Nov;15(11):935-45. doi: 10.1080/02699050110065295. PMID 11689092
- [Background] Simpson G, Tate R. Suicidality after traumatic brain injury: demographic, injury and clinical correlates. Psychol Med. 2002 May;32(4):687-97. doi: 10.1017/s0033291702005561. PMID 12102383
- [Background] Teasdale TW, Engberg AW. Suicide after traumatic brain injury: a population study. J Neurol Neurosurg Psychiatry. 2001 Oct;71(4):436-40. doi: 10.1136/jnnp.71.4.436. PMID 11561024
- [Background] Satz P, Forney DL, Zaucha K, Asarnow RR, Light R, McCleary C, Levin H, Kelly D, Bergsneider M, Hovda D, Martin N, Namerow N, Becker D. Depression, cognition, and functional correlates of recovery outcome after traumatic brain injury. Brain Inj. 1998 Jul;12(7):537-53. doi: 10.1080/026990598122313. PMID 9653518
- [Background] Deb S, Lyons I, Koutzoukis C, Ali I, McCarthy G. Rate of psychiatric illness 1 year after traumatic brain injury. Am J Psychiatry. 1999 Mar;156(3):374-8. doi: 10.1176/ajp.156.3.374. PMID 10080551
- [Background] Levin HS, Brown SA, Song JX, McCauley SR, Boake C, Contant CF, Goodman H, Kotrla KJ. Depression and posttraumatic stress disorder at three months after mild to moderate traumatic brain injury. J Clin Exp Neuropsychol. 2001 Dec;23(6):754-69. doi: 10.1076/jcen.23.6.754.1021. PMID 11910542
- [Background] Rapoport MJ, McCullagh S, Streiner D, Feinstein A. The clinical significance of major depression following mild traumatic brain injury. Psychosomatics. 2003 Jan-Feb;44(1):31-7. doi: 10.1176/appi.psy.44.1.31. PMID 12515835
- [Background] Franulic A, Carbonell CG, Pinto P, Sepulveda I. Psychosocial adjustment and employment outcome 2, 5 and 10 years after TBI. Brain Inj. 2004 Feb;18(2):119-29. doi: 10.1080/0269905031000149515. PMID 14660225
- [Background] Jorge RE, Robinson RG, Moser D, Tateno A, Crespo-Facorro B, Arndt S. Major depression following traumatic brain injury. Arch Gen Psychiatry. 2004 Jan;61(1):42-50. doi: 10.1001/archpsyc.61.1.42. PMID 14706943
- [Background] Rapoport MJ, McCullagh S, Shammi P, Feinstein A. Cognitive impairment associated with major depression following mild and moderate traumatic brain injury. J Neuropsychiatry Clin Neurosci. 2005 Winter;17(1):61-5. doi: 10.1176/jnp.17.1.61. PMID 15746484
- [Background] Trivedi MH, Greer TL, Grannemann BD, Chambliss HO, Jordan AN. Exercise as an augmentation strategy for treatment of major depression. J Psychiatr Pract. 2006 Jul;12(4):205-13. doi: 10.1097/00131746-200607000-00002. PMID 16883145
- [Background] Barbour KA, Edenfield TM, Blumenthal JA. Exercise as a treatment for depression and other psychiatric disorders: a review. J Cardiopulm Rehabil Prev. 2007 Nov-Dec;27(6):359-67. doi: 10.1097/01.HCR.0000300262.69645.95. PMID 18197069
- [Background] Cassilhas RC, Viana VA, Grassmann V, Santos RT, Santos RF, Tufik S, Mello MT. The impact of resistance exercise on the cognitive function of the elderly. Med Sci Sports Exerc. 2007 Aug;39(8):1401-7. doi: 10.1249/mss.0b013e318060111f. PMID 17762374
- [Background] Singh NA, Stavrinos TM, Scarbek Y, Galambos G, Liber C, Fiatarone Singh MA. A randomized controlled trial of high versus low intensity weight training versus general practitioner care for clinical depression in older adults. J Gerontol A Biol Sci Med Sci. 2005 Jun;60(6):768-76. doi: 10.1093/gerona/60.6.768. PMID 15983181
- [Background] Stein PN, Motta RW. Effects of aerobic and nonaerobic exercise on depression and self-concept. Percept Mot Skills. 1992 Feb;74(1):79-89. doi: 10.2466/pms.1992.74.1.79. PMID 1561044
- [Background] Doyne EJ, Ossip-Klein DJ, Bowman ED, Osborn KM, McDougall-Wilson IB, Neimeyer RA. Running versus weight lifting in the treatment of depression. J Consult Clin Psychol. 1987 Oct;55(5):748-54. doi: 10.1037//0022-006x.55.5.748. No abstract available. PMID 3454786
- [Background] Chen JK, Johnston KM, Petrides M, Ptito A. Neural substrates of symptoms of depression following concussion in male athletes with persisting postconcussion symptoms. Arch Gen Psychiatry. 2008 Jan;65(1):81-9. doi: 10.1001/archgenpsychiatry.2007.8. PMID 18180432
- [Background] Jorge RE, Acion L, Starkstein SE, Magnotta V. Hippocampal volume and mood disorders after traumatic brain injury. Biol Psychiatry. 2007 Aug 15;62(4):332-8. doi: 10.1016/j.biopsych.2006.07.024. Epub 2006 Nov 21. PMID 17123480
- [Background] Colcombe SJ, Erickson KI, Scalf PE, Kim JS, Prakash R, McAuley E, Elavsky S, Marquez DX, Hu L, Kramer AF. Aerobic exercise training increases brain volume in aging humans. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1166-70. doi: 10.1093/gerona/61.11.1166. PMID 17167157
- [Background] Pajonk FG, Wobrock T, Gruber O, Scherk H, Berner D, Kaizl I, Kierer A, Muller S, Oest M, Meyer T, Backens M, Schneider-Axmann T, Thornton AE, Honer WG, Falkai P. Hippocampal plasticity in response to exercise in schizophrenia. Arch Gen Psychiatry. 2010 Feb;67(2):133-43. doi: 10.1001/archgenpsychiatry.2009.193. PMID 20124113
- [Background] Langlois JA, Rutland-Brown W, Thomas KE. Traumatic brain injury in the United States: emergency department visits, hospitalizations, and deaths. Atlanta (GA): Centers for Disease Control and Prevention, Nation Center for Injury Prevention and Control. 2006.
- [Background] Thurman DJ, Alverson C, Dunn KA, Guerrero J, Sniezek JE. Traumatic brain injury in the United States: A public health perspective. J Head Trauma Rehabil. 1999 Dec;14(6):602-15. doi: 10.1097/00001199-199912000-00009. PMID 10671706
- [Background] Finkelstein E, Corso P, Miller T and associates. The Incidence and Economic Burden of Injuries in the United States. New York (NY): Oxford University Press. 2006.
- [Background] Mooney G, Speed J. The association between mild traumatic brain injury and psychiatric conditions. Brain Inj. 2001 Oct;15(10):865-77. doi: 10.1080/02699050110065286. PMID 11595083
- [Background] Underhill AT, Lobello SG, Stroud TP, Terry KS, Devivo MJ, Fine PR. Depression and life satisfaction in patients with traumatic brain injury: a longitudinal study. Brain Inj. 2003 Nov;17(11):973-82. doi: 10.1080/0269905031000110418. PMID 14514448
- [Background] Lee H, Kim SW, Kim JM, Shin IS, Yang SJ, Yoon JS. Comparing effects of methylphenidate, sertraline and placebo on neuropsychiatric sequelae in patients with traumatic brain injury. Hum Psychopharmacol. 2005 Mar;20(2):97-104. doi: 10.1002/hup.668. PMID 15641125
- [Background] Olfson M, Marcus SC. National patterns in antidepressant medication treatment. Arch Gen Psychiatry. 2009 Aug;66(8):848-56. doi: 10.1001/archgenpsychiatry.2009.81. PMID 19652124
- [Background] Fann JR, Hart T, Schomer KG. Treatment for depression after traumatic brain injury: a systematic review. J Neurotrauma. 2009 Dec;26(12):2383-402. doi: 10.1089/neu.2009.1091. PMID 19698070
- [Background] Topolovec-Vranic J, Cullen N, Michalak A, Ouchterlony D, Bhalerao S, Masanic C, Cusimano MD. Evaluation of an online cognitive behavioural therapy program by patients with traumatic brain injury and depression. Brain Inj. 2010;24(5):762-72. doi: 10.3109/02699051003709599. PMID 20370383
- [Background] Bombardier CH, Bell KR, Temkin NR, Fann JR, Hoffman J, Dikmen S. The efficacy of a scheduled telephone intervention for ameliorating depressive symptoms during the first year after traumatic brain injury. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):230-8. doi: 10.1097/HTR.0b013e3181ad65f0. PMID 19625862
- [Background] Trivedi MH, Greer TL, Grannemann BD, Church TS, Galper DI, Sunderajan P, Wisniewski SR, Chambliss HO, Jordan AN, Finley C, Carmody TI. TREAD: TReatment with Exercise Augmentation for Depression: study rationale and design. Clin Trials. 2006;3(3):291-305. doi: 10.1191/1740774506cn151oa. PMID 16895046
- [Background] Singh NA, Clements KM, Singh MA. The efficacy of exercise as a long-term antidepressant in elderly subjects: a randomized, controlled trial. J Gerontol A Biol Sci Med Sci. 2001 Aug;56(8):M497-504. doi: 10.1093/gerona/56.8.m497. PMID 11487602
- [Background] Gordon WA, Sliwinski M, Echo J, McLoughlin M, Sheerer MS, Meili TE. The benefits of exercise in individuals with traumatic brain injury: a retrospective study. J Head Trauma Rehabil. 1998 Aug;13(4):58-67. doi: 10.1097/00001199-199808000-00006. PMID 9651240
- [Background] Driver S, Ede A. Impact of physical activity on mood after TBI. Brain Inj. 2009 Mar;23(3):203-12. doi: 10.1080/02699050802695574. PMID 19205956
- [Background] Maletic V, Robinson M, Oakes T, Iyengar S, Ball SG, Russell J. Neurobiology of depression: an integrated view of key findings. Int J Clin Pract. 2007 Dec;61(12):2030-40. doi: 10.1111/j.1742-1241.2007.01602.x. Epub 2007 Oct 17. PMID 17944926
- [Background] McEwen BS. Glucocorticoids, depression, and mood disorders: structural remodeling in the brain. Metabolism. 2005 May;54(5 Suppl 1):20-3. doi: 10.1016/j.metabol.2005.01.008. PMID 15877308
- [Background] Lee AL, Ogle WO, Sapolsky RM. Stress and depression: possible links to neuron death in the hippocampus. Bipolar Disord. 2002 Apr;4(2):117-28. doi: 10.1034/j.1399-5618.2002.01144.x. PMID 12071509
- [Background] Aihara M, Ida I, Yuuki N, Oshima A, Kumano H, Takahashi K, Fukuda M, Oriuchi N, Endo K, Matsuda H, Mikuni M. HPA axis dysfunction in unmedicated major depressive disorder and its normalization by pharmacotherapy correlates with alteration of neural activity in prefrontal cortex and limbic/paralimbic regions. Psychiatry Res. 2007 Aug 15;155(3):245-56. doi: 10.1016/j.pscychresns.2006.11.002. Epub 2007 Jun 22. PMID 17587554
- [Background] Starkman MN, Gebarski SS, Berent S, Schteingart DE. Hippocampal formation volume, memory dysfunction, and cortisol levels in patients with Cushing's syndrome. Biol Psychiatry. 1992 Nov 1;32(9):756-65. doi: 10.1016/0006-3223(92)90079-f. PMID 1450290
- [Background] Van Den Eede F, Van den Bossche B, Hulstijn W, Sabbe BG, Cosyns P, Claes SJ. Combined dexamethasone/CRF test in remitted outpatients with recurrent major depressive disorder. J Affect Disord. 2006 Jul;93(1-3):259-63. doi: 10.1016/j.jad.2006.03.020. Epub 2006 May 4. PMID 16677715
- [Background] Holsboer F. The rationale for corticotropin-releasing hormone receptor (CRH-R) antagonists to treat depression and anxiety. J Psychiatr Res. 1999 May-Jun;33(3):181-214. doi: 10.1016/s0022-3956(98)90056-5. PMID 10367986
- [Background] Holsboer F. The corticosteroid receptor hypothesis of depression. Neuropsychopharmacology. 2000 Nov;23(5):477-501. doi: 10.1016/S0893-133X(00)00159-7. PMID 11027914
- [Background] Ghigo E, Masel B, Aimaretti G, Leon-Carrion J, Casanueva FF, Dominguez-Morales MR, Elovic E, Perrone K, Stalla G, Thompson C, Urban R. Consensus guidelines on screening for hypopituitarism following traumatic brain injury. Brain Inj. 2005 Aug 20;19(9):711-24. doi: 10.1080/02699050400025315. PMID 16195185
- [Background] Fedoroff JP, Starkstein SE, Forrester AW, Geisler FH, Jorge RE, Arndt SV, Robinson RG. Depression in patients with acute traumatic brain injury. Am J Psychiatry. 1992 Jul;149(7):918-23. doi: 10.1176/ajp.149.7.918. PMID 1609872
- [Background] Jorge R, Robinson RG. Mood disorders following traumatic brain injury. NeuroRehabilitation. 2002;17(4):311-24. No abstract available. PMID 12547979
- [Background] Ernst C, Olson AK, Pinel JP, Lam RW, Christie BR. Antidepressant effects of exercise: evidence for an adult-neurogenesis hypothesis? J Psychiatry Neurosci. 2006 Mar;31(2):84-92. PMID 16575423
- [Background] Eriksson PS, Perfilieva E, Bjork-Eriksson T, Alborn AM, Nordborg C, Peterson DA, Gage FH. Neurogenesis in the adult human hippocampus. Nat Med. 1998 Nov;4(11):1313-7. doi: 10.1038/3305. PMID 9809557
- [Background] Koolschijn PC, van Haren NE, Lensvelt-Mulders GJ, Hulshoff Pol HE, Kahn RS. Brain volume abnormalities in major depressive disorder: a meta-analysis of magnetic resonance imaging studies. Hum Brain Mapp. 2009 Nov;30(11):3719-35. doi: 10.1002/hbm.20801. PMID 19441021
- [Background] Videbech P, Ravnkilde B. Hippocampal volume and depression: a meta-analysis of MRI studies. Am J Psychiatry. 2004 Nov;161(11):1957-66. doi: 10.1176/appi.ajp.161.11.1957. PMID 15514393
- [Background] Yucel K, McKinnon MC, Chahal R, Taylor VH, Macdonald K, Joffe R, MacQueen GM. Anterior cingulate volumes in never-treated patients with major depressive disorder. Neuropsychopharmacology. 2008 Dec;33(13):3157-63. doi: 10.1038/npp.2008.40. Epub 2008 Mar 26. PMID 18368034
- [Background] Mak AK, Wong MM, Han SH, Lee TM. Gray matter reduction associated with emotion regulation in female outpatients with major depressive disorder: a voxel-based morphometry study. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Oct 1;33(7):1184-90. doi: 10.1016/j.pnpbp.2009.06.025. Epub 2009 Jul 19. PMID 19596037
- [Background] Sapolsky RM. Glucocorticoids and hippocampal atrophy in neuropsychiatric disorders. Arch Gen Psychiatry. 2000 Oct;57(10):925-35. doi: 10.1001/archpsyc.57.10.925. PMID 11015810
- [Background] Czeh B, Lucassen PJ. What causes the hippocampal volume decrease in depression? Are neurogenesis, glial changes and apoptosis implicated? Eur Arch Psychiatry Clin Neurosci. 2007 Aug;257(5):250-60. doi: 10.1007/s00406-007-0728-0. PMID 17401728
- [Background] Henn FA, Vollmayr B. Neurogenesis and depression: etiology or epiphenomenon? Biol Psychiatry. 2004 Aug 1;56(3):146-50. doi: 10.1016/j.biopsych.2004.04.011. PMID 15271582
- [Background] Duman RS. Depression: a case of neuronal life and death? Biol Psychiatry. 2004 Aug 1;56(3):140-5. doi: 10.1016/j.biopsych.2004.02.033. PMID 15271581
- [Background] Cotter DR, Pariante CM, Everall IP. Glial cell abnormalities in major psychiatric disorders: the evidence and implications. Brain Res Bull. 2001 Jul 15;55(5):585-95. doi: 10.1016/s0361-9230(01)00527-5. PMID 11576755
- [Background] Rajkowska G. Cell pathology in mood disorders. Semin Clin Neuropsychiatry. 2002 Oct;7(4):281-92. doi: 10.1053/scnp.2002.35228. PMID 12382210
- [Background] van Praag H, Shubert T, Zhao C, Gage FH. Exercise enhances learning and hippocampal neurogenesis in aged mice. J Neurosci. 2005 Sep 21;25(38):8680-5. doi: 10.1523/JNEUROSCI.1731-05.2005. PMID 16177036
- [Background] van Praag H, Christie BR, Sejnowski TJ, Gage FH. Running enhances neurogenesis, learning, and long-term potentiation in mice. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13427-31. doi: 10.1073/pnas.96.23.13427. PMID 10557337
- [Background] van Praag H, Kempermann G, Gage FH. Running increases cell proliferation and neurogenesis in the adult mouse dentate gyrus. Nat Neurosci. 1999 Mar;2(3):266-70. doi: 10.1038/6368. PMID 10195220
- [Background] Erickson KI, Prakash RS, Voss MW, Chaddock L, Hu L, Morris KS, White SM, Wojcicki TR, McAuley E, Kramer AF. Aerobic fitness is associated with hippocampal volume in elderly humans. Hippocampus. 2009 Oct;19(10):1030-9. doi: 10.1002/hipo.20547. PMID 19123237
- [Background] Palmer TD, Willhoite AR, Gage FH. Vascular niche for adult hippocampal neurogenesis. J Comp Neurol. 2000 Oct 2;425(4):479-94. doi: 10.1002/1096-9861(20001002)425:43.0.co;2-3. PMID 10975875
- [Background] Louissaint A Jr, Rao S, Leventhal C, Goldman SA. Coordinated interaction of neurogenesis and angiogenesis in the adult songbird brain. Neuron. 2002 Jun 13;34(6):945-60. doi: 10.1016/s0896-6273(02)00722-5. PMID 12086642
- [Background] Pereira AC, Huddleston DE, Brickman AM, Sosunov AA, Hen R, McKhann GM, Sloan R, Gage FH, Brown TR, Small SA. An in vivo correlate of exercise-induced neurogenesis in the adult dentate gyrus. Proc Natl Acad Sci U S A. 2007 Mar 27;104(13):5638-43. doi: 10.1073/pnas.0611721104. Epub 2007 Mar 20. PMID 17374720
- [Background] Warner-Schmidt JL, Duman RS. VEGF as a potential target for therapeutic intervention in depression. Curr Opin Pharmacol. 2008 Feb;8(1):14-9. doi: 10.1016/j.coph.2007.10.013. Epub 2007 Dec 3. PMID 18061540
- [Background] Mira H, Andreu Z, Suh H, Lie DC, Jessberger S, Consiglio A, San Emeterio J, Hortiguela R, Marques-Torrejon MA, Nakashima K, Colak D, Gotz M, Farinas I, Gage FH. Signaling through BMPR-IA regulates quiescence and long-term activity of neural stem cells in the adult hippocampus. Cell Stem Cell. 2010 Jul 2;7(1):78-89. doi: 10.1016/j.stem.2010.04.016. PMID 20621052
- [Background] Piser TM. Linking the cytokine and neurocircuitry hypotheses of depression: a translational framework for discovery and development of novel anti-depressants. Brain Behav Immun. 2010 May;24(4):515-24. doi: 10.1016/j.bbi.2010.02.006. Epub 2010 Mar 1. PMID 20193757
- [Background] Gervasoni N, Aubry JM, Bondolfi G, Osiek C, Schwald M, Bertschy G, Karege F. Partial normalization of serum brain-derived neurotrophic factor in remitted patients after a major depressive episode. Neuropsychobiology. 2005;51(4):234-8. doi: 10.1159/000085725. Epub 2005 May 12. PMID 15897674
- [Background] Aydemir O, Deveci A, Taneli F. The effect of chronic antidepressant treatment on serum brain-derived neurotrophic factor levels in depressed patients: a preliminary study. Prog Neuropsychopharmacol Biol Psychiatry. 2005 Feb;29(2):261-5. doi: 10.1016/j.pnpbp.2004.11.009. Epub 2004 Dec 23. PMID 15694233
- [Background] Shimizu E, Hashimoto K, Okamura N, Koike K, Komatsu N, Kumakiri C, Nakazato M, Watanabe H, Shinoda N, Okada S, Iyo M. Alterations of serum levels of brain-derived neurotrophic factor (BDNF) in depressed patients with or without antidepressants. Biol Psychiatry. 2003 Jul 1;54(1):70-5. doi: 10.1016/s0006-3223(03)00181-1. PMID 12842310
- [Background] Gonul AS, Akdeniz F, Taneli F, Donat O, Eker C, Vahip S. Effect of treatment on serum brain-derived neurotrophic factor levels in depressed patients. Eur Arch Psychiatry Clin Neurosci. 2005 Dec;255(6):381-6. doi: 10.1007/s00406-005-0578-6. Epub 2005 Apr 6. PMID 15809771
- [Background] Nibuya M, Morinobu S, Duman RS. Regulation of BDNF and trkB mRNA in rat brain by chronic electroconvulsive seizure and antidepressant drug treatments. J Neurosci. 1995 Nov;15(11):7539-47. doi: 10.1523/JNEUROSCI.15-11-07539.1995. PMID 7472505
- [Background] Warner-Schmidt JL, Duman RS. VEGF is an essential mediator of the neurogenic and behavioral actions of antidepressants. Proc Natl Acad Sci U S A. 2007 Mar 13;104(11):4647-52. doi: 10.1073/pnas.0610282104. Epub 2007 Mar 5. PMID 17360578
- [Background] Sen S, Duman R, Sanacora G. Serum brain-derived neurotrophic factor, depression, and antidepressant medications: meta-analyses and implications. Biol Psychiatry. 2008 Sep 15;64(6):527-32. doi: 10.1016/j.biopsych.2008.05.005. Epub 2008 Jun 24. PMID 18571629
- [Background] Shirayama Y, Chen AC, Nakagawa S, Russell DS, Duman RS. Brain-derived neurotrophic factor produces antidepressant effects in behavioral models of depression. J Neurosci. 2002 Apr 15;22(8):3251-61. doi: 10.1523/JNEUROSCI.22-08-03251.2002. PMID 11943826
- [Background] Siuciak JA, Lewis DR, Wiegand SJ, Lindsay RM. Antidepressant-like effect of brain-derived neurotrophic factor (BDNF). Pharmacol Biochem Behav. 1997 Jan;56(1):131-7. doi: 10.1016/S0091-3057(96)00169-4. PMID 8981620
- [Background] Koponen E, Rantamaki T, Voikar V, Saarelainen T, MacDonald E, Castren E. Enhanced BDNF signaling is associated with an antidepressant-like behavioral response and changes in brain monoamines. Cell Mol Neurobiol. 2005 Sep;25(6):973-80. doi: 10.1007/s10571-005-8468-z. PMID 16392030
- [Background] Hoshaw BA, Malberg JE, Lucki I. Central administration of IGF-I and BDNF leads to long-lasting antidepressant-like effects. Brain Res. 2005 Mar 10;1037(1-2):204-8. doi: 10.1016/j.brainres.2005.01.007. PMID 15777771
- [Background] Kiraly MA, Kiraly SJ. The effect of exercise on hippocampal integrity: review of recent research. Int J Psychiatry Med. 2005;35(1):75-89. doi: 10.2190/HX7L-4B40-PQNY-2A4P. PMID 15977946
- [Background] Vaynman S, Ying Z, Gomez-Pinilla F. Hippocampal BDNF mediates the efficacy of exercise on synaptic plasticity and cognition. Eur J Neurosci. 2004 Nov;20(10):2580-90. doi: 10.1111/j.1460-9568.2004.03720.x. PMID 15548201
- [Background] Fabel K, Fabel K, Tam B, Kaufer D, Baiker A, Simmons N, Kuo CJ, Palmer TD. VEGF is necessary for exercise-induced adult hippocampal neurogenesis. Eur J Neurosci. 2003 Nov;18(10):2803-12. doi: 10.1111/j.1460-9568.2003.03041.x. PMID 14656329
- [Background] Mossberg KA, Amonette WE, Masel BE. Endurance training and cardiorespiratory conditioning after traumatic brain injury. J Head Trauma Rehabil. 2010 May-Jun;25(3):173-83. doi: 10.1097/HTR.0b013e3181dc98ff. PMID 20473091
- [Background] Beck, Aaron T., Robert A. Steer, and Gregory K. Brown. BDI-II, Beck Depression Inventory: Manual. San Antonio, Tex: Psychological Corp, 1996
- [Background] Jezierski MK, Sohrabji F. Region- and peptide-specific regulation of the neurotrophins by estrogen. Brain Res Mol Brain Res. 2000 Dec 28;85(1-2):77-84. doi: 10.1016/s0169-328x(00)00244-8. PMID 11146109
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Background] Borg, GAV. Physical Performance and Perceived Exertion. Lund, Sweden: Gleerup.
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Dale AM, Sereno MI. Improved Localizadon of Cortical Activity by Combining EEG and MEG with MRI Cortical Surface Reconstruction: A Linear Approach. J Cogn Neurosci. 1993 Spring;5(2):162-76. doi: 10.1162/jocn.1993.5.2.162. PMID 23972151
- [Background] Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):11050-5. doi: 10.1073/pnas.200033797. PMID 10984517
- [Background] Fischl B, Liu A, Dale AM. Automated manifold surgery: constructing geometrically accurate and topologically correct models of the human cerebral cortex. IEEE Trans Med Imaging. 2001 Jan;20(1):70-80. doi: 10.1109/42.906426. PMID 11293693
- [Background] Fischl B, Salat DH, Busa E, Albert M, Dieterich M, Haselgrove C, van der Kouwe A, Killiany R, Kennedy D, Klaveness S, Montillo A, Makris N, Rosen B, Dale AM. Whole brain segmentation: automated labeling of neuroanatomical structures in the human brain. Neuron. 2002 Jan 31;33(3):341-55. doi: 10.1016/s0896-6273(02)00569-x. PMID 11832223
- [Background] Fischl B, Salat DH, van der Kouwe AJ, Makris N, Segonne F, Quinn BT, Dale AM. Sequence-independent segmentation of magnetic resonance images. Neuroimage. 2004;23 Suppl 1:S69-84. doi: 10.1016/j.neuroimage.2004.07.016. PMID 15501102
- [Background] Fischl B, Sereno MI, Dale AM. Cortical surface-based analysis. II: Inflation, flattening, and a surface-based coordinate system. Neuroimage. 1999 Feb;9(2):195-207. doi: 10.1006/nimg.1998.0396. PMID 9931269
- [Background] Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. Hum Brain Mapp. 1999;8(4):272-84. doi: 10.1002/(sici)1097-0193(1999)8:43.0.co;2-4. PMID 10619420
- [Background] Fischl B, van der Kouwe A, Destrieux C, Halgren E, Segonne F, Salat DH, Busa E, Seidman LJ, Goldstein J, Kennedy D, Caviness V, Makris N, Rosen B, Dale AM. Automatically parcellating the human cerebral cortex. Cereb Cortex. 2004 Jan;14(1):11-22. doi: 10.1093/cercor/bhg087. PMID 14654453
- [Background] Han X, Jovicich J, Salat D, van der Kouwe A, Quinn B, Czanner S, Busa E, Pacheco J, Albert M, Killiany R, Maguire P, Rosas D, Makris N, Dale A, Dickerson B, Fischl B. Reliability of MRI-derived measurements of human cerebral cortical thickness: the effects of field strength, scanner upgrade and manufacturer. Neuroimage. 2006 Aug 1;32(1):180-94. doi: 10.1016/j.neuroimage.2006.02.051. Epub 2006 May 2. PMID 16651008
- [Background] Jovicich J, Czanner S, Greve D, Haley E, van der Kouwe A, Gollub R, Kennedy D, Schmitt F, Brown G, Macfall J, Fischl B, Dale A. Reliability in multi-site structural MRI studies: effects of gradient non-linearity correction on phantom and human data. Neuroimage. 2006 Apr 1;30(2):436-43. doi: 10.1016/j.neuroimage.2005.09.046. Epub 2005 Nov 21. PMID 16300968
- [Background] Segonne F, Dale AM, Busa E, Glessner M, Salat D, Hahn HK, Fischl B. A hybrid approach to the skull stripping problem in MRI. Neuroimage. 2004 Jul;22(3):1060-75. doi: 10.1016/j.neuroimage.2004.03.032. PMID 15219578
- [Background] Dale AM, Fischl B, Sereno MI. Cortical surface-based analysis. I. Segmentation and surface reconstruction. Neuroimage. 1999 Feb;9(2):179-94. doi: 10.1006/nimg.1998.0395. PMID 9931268
- [Background] Salat DH, Buckner RL, Snyder AZ, Greve DN, Desikan RS, Busa E, Morris JC, Dale AM, Fischl B. Thinning of the cerebral cortex in aging. Cereb Cortex. 2004 Jul;14(7):721-30. doi: 10.1093/cercor/bhh032. Epub 2004 Mar 28. PMID 15054051
- [Background] Kuperberg GR, Broome MR, McGuire PK, David AS, Eddy M, Ozawa F, Goff D, West WC, Williams SC, van der Kouwe AJ, Salat DH, Dale AM, Fischl B. Regionally localized thinning of the cerebral cortex in schizophrenia. Arch Gen Psychiatry. 2003 Sep;60(9):878-88. doi: 10.1001/archpsyc.60.9.878. PMID 12963669
- [Background] Rosas HD, Liu AK, Hersch S, Glessner M, Ferrante RJ, Salat DH, van der Kouwe A, Jenkins BG, Dale AM, Fischl B. Regional and progressive thinning of the cortical ribbon in Huntington's disease. Neurology. 2002 Mar 12;58(5):695-701. doi: 10.1212/wnl.58.5.695. PMID 11889230
- [Background] Kashihara K, Maruyama T, Murota M, Nakahara Y. Positive effects of acute and moderate physical exercise on cognitive function. J Physiol Anthropol. 2009 Jun;28(4):155-64. doi: 10.2114/jpa2.28.155. PMID 19652447
- [Background] McDermott LM, Ebmeier KP. A meta-analysis of depression severity and cognitive function. J Affect Disord. 2009 Dec;119(1-3):1-8. doi: 10.1016/j.jad.2009.04.022. Epub 2009 May 9. PMID 19428120
- [Background] Bagiella E, Novack TA, Ansel B, Diaz-Arrastia R, Dikmen S, Hart T, Temkin N. Measuring outcome in traumatic brain injury treatment trials: recommendations from the traumatic brain injury clinical trials network. J Head Trauma Rehabil. 2010 Sep-Oct;25(5):375-82. doi: 10.1097/HTR.0b013e3181d27fe3. PMID 20216459
- [Background] Benton AL, Hamsher KD, Sivan AB. Multilingual Aphasia Examination. Manual of instructions. AJA Associates, Iowa City. 2000.
- [Background] Reitan RM, Wolfson D. The Halstead-Reitan neuropsychological test battery: Theory and clinical interpretation. Neuropsychology Press, Tucson, AZ. 1993.
- [Background] Reitan RM Trail Making Test. Manual for administration and scoring. Reitan Neuropsychology Laboratory, Tucson, AZ. 1992.
- [Background] Dodrill CB. A neuropsychological battery for epilepsy. Epilepsia. 1978 Dec;19(6):611-23. doi: 10.1111/j.1528-1157.1978.tb05041.x. PMID 738230
- [Background] Wechsler D. Wechsler Adult Intelligence Scale (WAIS-III). The Psychological Corporation, San Antonio, TX. 1997.
- [Background] Delis DCK, Joel H, Kaplan E, Ober BA. California Verbal Learning Test. PsychCorp, A brand of Harcourt Assessment, Inc. 2000.
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Noble BJ, Borg GA, Jacobs I, Ceci R, Kaiser P. A category-ratio perceived exertion scale: relationship to blood and muscle lactates and heart rate. Med Sci Sports Exerc. 1983;15(6):523-8. PMID 6656563
- [Background] Rappaport M, Hall KM, Hopkins K, Belleza T, Cope DN. Disability rating scale for severe head trauma: coma to community. Arch Phys Med Rehabil. 1982 Mar;63(3):118-23. PMID 7073452
- [Background] Gouvier WD, Blanton PD, LaPorte KK, Nepomuceno C. Reliability and validity of the Disability Rating Scale and the Levels of Cognitive Functioning Scale in monitoring recovery from severe head injury. Arch Phys Med Rehabil. 1987 Feb;68(2):94-7. PMID 3813863
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Chew E, Zafonte RD. Pharmacological management of neurobehavioral disorders following traumatic brain injury--a state-of-the-art review. J Rehabil Res Dev. 2009;46(6):851-79. doi: 10.1682/jrrd.2008.09.0120. PMID 20104408
- [Background] Neurobehavioral Guidelines Working Group; Warden DL, Gordon B, McAllister TW, Silver JM, Barth JT, Bruns J, Drake A, Gentry T, Jagoda A, Katz DI, Kraus J, Labbate LA, Ryan LM, Sparling MB, Walters B, Whyte J, Zapata A, Zitnay G. Guidelines for the pharmacologic treatment of neurobehavioral sequelae of traumatic brain injury. J Neurotrauma. 2006 Oct;23(10):1468-501. doi: 10.1089/neu.2006.23.1468. PMID 17020483
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences, (revised edition). New York. NY: Academic Press, 1977
- See also: Arhinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts freely available online — http://surfer.nmr.mgh.harvard.edu